CLINICAL TRIAL: NCT05504200
Title: Promoting Restoration of Function of Co-ordinated Bladder Storage and Voiding Following Spinal Cord Injury by Combination of Transcutaneous Spinal Cord Stimulation and Bladder & Pelvic Floor Muscle Training Training
Brief Title: Transcutaneous Spinal Cord Stimulation With Bladder and Pelvic Floor Muscle Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RNOH RIC (Other)
Collaborators: International Spinal Research Trust (Other)
Responsible Party: Sponsor-Investigator, RNOH RIC, Head of Research and Innovation, Royal National Orthopaedic Hospital NHS Trust
Organization: Royal National Orthopaedic Hospital NHS Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 304762
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal cord stimulation; Pelvic floor physiotherapy; Incontinence; Bladder overactivity; Neurogenic detrusor overactivity
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bladder and Pelvic Floor Muscle Training (Experimental): Participants randomised to the intervention group will complete an 8-week bladder and PFMT programme, both at the LSCIC and at home. They will be invited to 3 face-to-face follow up appointments over the 8-weeks, where they will meet with a physiotherapist to check their technique and monitor their progress. At home participants will receive a daily text reminder to complete their PFM training, they will also receive a weekly phone call from a member of the research team who will check how they are managing and whether they have any questions. At the end of the programme, participants will be asked to repeat the questionnaires and have their pelvic floor re-assessed. Following this, they will complete the urodynamic investigation with tSCS.
  Interventions: Other: Bladder and Pelvic Floor Muscle Training
- Control (No Intervention): Participants randomised to the control group will continue with their usual care for 8-weeks. They will return to repeat their baseline questionnaires and have their pelvic floor re-assessed. Finally, they will complete tSCS bladder filling and emptying cycles with urodynamics.

INTERVENTIONS:
Other: Bladder and Pelvic Floor Muscle Training — The intervention group will receive 8-weeks of at home PFMT, this will include 3 face-to-face visits, daily text reminders, and a weekly phone call.
  Arms: Bladder and Pelvic Floor Muscle Training

SUMMARY:
Spinal Cord Injury (SCI) disrupts signals between the brain and the rest of the body, this includes signals needed to control the bladder and bowels. Spinal cord stimulation (SCS) (electrical stimulation through electrodes placed on the skin over the spine) has shown potential to improve bladder function. Additionally pelvic floor muscle training (PFMT), has been shown to help control bladder overactivity and reduce incontinence in people with a SCI.

This study will investigate PFMT with SCS, and its effects on restoring bladder function, and continence. We aim to recruit 25 participants. Those eligible will be patients from the London Spinal Cord Injury Centre with a supra-sacral SCI (>6 months post-injury), aged 16 years old and above.

DETAILED DESCRIPTION:
The first five participants who volunteer will be invited to complete 'SCS optimisation'. Testing different SCS electrode positions and stimulation parameters with pelvic floor exercises and during urodynamics (measurement of pressure changes during filling and emptying of the bladder).

For the main study, all participants will complete baseline assessments (week 1) which include: bladder, bowel, sexual function, and quality of life questionnaires, a pelvic floor assessment, and urodynamics. Assessments will be repeated at week 8, and week 14.

After baseline assessments, participants will be randomly allocated to one of two groups. The intervention group will receive 8-weeks of at home PFMT, this will include 3 face-to-face visits, daily text reminders, and a weekly phone call. The control group will continue with usual care for 8-weeks.

At the end of the 8-weeks, all participants will be re-assessed, and will then complete a single session of SCS with urodynamics. Participants will return for their final assessment 6-weeks later (week 14). Participants allocated to the control group will be offered PFMT at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Supra-sacral spinal cord injury over 6 months ago
* Previous urodynamics and management by the Neuro-urology Consultants
* Proven NDO from latest urodynamics

Exclusion Criteria:

* Participants under 16 years of age
* Non-stable SCI or metastatic cord disease
* Intra-detrusor botulinum toxin injections in previous 6 months
* Bladder infection on day of investigation
* Pregnant or trying for a baby (females)
* Cardiac pacemaker, bladder stimulator or baclofen pump in situ
* Metal work at thoraco-lumbar level of stimulation
* Poorly controlled Autonomic Dysreflexia
* Currently involved in a clinical trial
* Previous surgical intervention on bladder/sphincters
* Active sepsis
* Poorly controlled epilepsy. Acceptable where epilepsy is controlled by drugs or there have been no fits experienced for a reasonable period
* Patients with a cancerous tumour in the area of the electrical stimulation
* Patients without the capacity to consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2023-09-04 (Actual); Study Completion 2023-09-04 (Actual)

PRIMARY OUTCOMES:
Change in maximum cystometric capacity (MCC) from baseline to follow up | Week 1, 8 and 14
  Bladder capacity from Cystometrogram/Urodynamic procedures (ml)
Change in maximum detrusor pressure during voiding (MDPvoid) from baseline to follow up | Week 1, 8 and 14
  Voiding detrusor pressure measured from Cystometrogram/Urodynamic procedures (cmH20)
Change in bladder voiding efficiency from baseline to follow up | Week 1, 8 and 14
  Bladder voiding efficiency measured from Cystometrogram/Urodynamic procedures, [[volume voided/volume voided+post void residual)*100] (%)

SECONDARY OUTCOMES:
Pelvic Floor Oxford Grading Score | Week 1, 8 and 14
  Measure of pelvic floor muscle strength, graded 0-5
The Neurogenic Bladder Symptom Score (NBSS) | Week 1, 8 and 14
  Validated 24-item questionnaire, three domains: incontinence, storage and voiding, consequences (score 0-28)
Neurogenic Bowel Dysfunction Score (NBDS) | Week 1, 8 and 14
  Bowel dysfunction questionnaire, includes questions on bowel symptoms, medication, and incontinence (score 0-47)
Arizona Sexual Experiences Scale (ASEX) | Week 1, 8 and 14
  Five-item rating scale measuring sex drive, arousal, vaginal lubrication/penile erection, ability to reach orgasm, and satisfaction from orgasm (Score 3-30)
Quality of Life Questionnaire EQ-5D-5L | Week 1, 8 and 14
  Five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Scoring 1-5 on each dimension, and a VAS scale of overall health 0-100.
The Qualiveen Questionnaire | Week 1, 8 and 14
  30-item questionnaire, with health-related quality of life questions specific to individuals with neurogenic urinary dysfunction. Total score is mean of eight scores: bother with limitations, fears, feelings, and frequency of limitations.
Electromyography (EMG) of resting tone and maximum voluntary pelvic floor contraction | Week 1, 8 and 14
  Use of vaginal/anal probe to capture resting tone and maximum voluntary pelvic floor contraction (mV)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Lee, Principal Investigator — Royal National Orthopaedic Hospital
Locations (1):
- Royal National Orthopaedic Hospital, Stanmore, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herrity AN, Aslan SC, Mesbah S, Siu R, Kalvakuri K, Ugiliweneza B, Mohamed A, Hubscher CH, Harkema SJ. Targeting bladder function with network-specific epidural stimulation after chronic spinal cord injury. Sci Rep. 2022 Jul 1;12(1):11179. doi: 10.1038/s41598-022-15315-2. PMID 35778466
- [Background] Gad PN, Kreydin E, Zhong H, Latack K, Edgerton VR. Non-invasive Neuromodulation of Spinal Cord Restores Lower Urinary Tract Function After Paralysis. Front Neurosci. 2018 Jun 29;12:432. doi: 10.3389/fnins.2018.00432. eCollection 2018. PMID 30008661
- [Background] Doherty S, Vanhoestenberghe A, Duffell L, Hamid R, Knight S. A Urodynamic Comparison of Neural Targets for Transcutaneous Electrical Stimulation to Acutely Suppress Detrusor Contractions Following Spinal Cord Injury. Front Neurosci. 2019 Dec 17;13:1360. doi: 10.3389/fnins.2019.01360. eCollection 2019. PMID 31956301
- [Background] Doherty SP, Vanhoestenberghe A, Duffell LD, Hamid R, Knight SL. Ambulatory urodynamic monitoring assessment of dorsal genital nerve stimulation for suppression of involuntary detrusor contractions following spinal cord injury: a pilot study. Spinal Cord Ser Cases. 2020 Apr 30;6(1):30. doi: 10.1038/s41394-020-0279-4. PMID 32355163
- [Background] Xu L, Fu C, Zhang Q, Xiong F, Peng L, Liang Z, Chen L, He C, Wei Q. Efficacy of biofeedback, repetitive transcranial magnetic stimulation and pelvic floor muscle training for female neurogenic bladder dysfunction after spinal cord injury: a study protocol for a randomised controlled trial. BMJ Open. 2020 Aug 5;10(8):e034582. doi: 10.1136/bmjopen-2019-034582. PMID 32759239
- [Background] Elmelund M, Biering-Sorensen F, Due U, Klarskov N. The effect of pelvic floor muscle training and intravaginal electrical stimulation on urinary incontinence in women with incomplete spinal cord injury: an investigator-blinded parallel randomized clinical trial. Int Urogynecol J. 2018 Nov;29(11):1597-1606. doi: 10.1007/s00192-018-3630-6. Epub 2018 Mar 24. PMID 29574482
- [Background] Vasquez N, Knight SL, Susser J, Gall A, Ellaway PH, Craggs MD. Pelvic floor muscle training in spinal cord injury and its impact on neurogenic detrusor over-activity and incontinence. Spinal Cord. 2015 Dec;53(12):887-9. doi: 10.1038/sc.2015.121. Epub 2015 Aug 4. PMID 26238317